CLINICAL TRIAL: NCT06263179
Title: Feasibility of Aerobic Exercise for Recovery From Work-related Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jacob I. McPherson, Clinical Assistant Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007706; UL1TR001412 (NIH)
Record Dates: First submitted 2024-01-29; First posted 2024-02-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Target Heartrate Aerobic Exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Target Heartrate Aerobic Exercise (THRAE) (Experimental): Participants will be asked to complete the Buffalo Concussion Treadmill Test (BCTT), a safe graded exercise test that is used to identify concussion-related exertion intolerance. Participants will wear a heart rate (HR) monitor for the collection of continuous HR data. The test is stopped when a participant's symptoms increase subjectively by an intensity of 3 points or more from the pre-exercise value on a scale from 0-10, or they report being physically exhausted. Their HR at the time of test termination constitutes the HR threshold (HRt). An individualized THRAE program will be prescribed based on 80% of the HRt on the BCTT. Participants will be given a Polar HR monitor to wear while performing their THRAE prescription, which will be performed at home for 20 minutes, 4-5 days per week, for 6 weeks or until medically cleared from their concussion.
  Interventions: Behavioral: Target Heartrate Aerobic Exercise

INTERVENTIONS:
Behavioral: Target Heartrate Aerobic Exercise — Exercise program

SUMMARY:
There is a lot of research on how to treat people with sport-related concussion. There has not been a lot of research on the treatment of injured workers with concussion. An exercise program has been developed for people with sport-related concussion. It is suspected that this program may be helpful for injured workers with concussion too. This study will test the effect of this exercise in injured workers with concussion.

DETAILED DESCRIPTION:
Participants who are diagnosed with a concussion and agree to participant in the study will complete a demographics form and other relevant questionnaires. They will then perform a graded exertion test (the Buffalo Concussion Treadmill Test [BCTT]) at the clinic, this takes approximately 15 minutes. Participants will then be prescribed the individualized THRAE based on the results from the BCTT and will be sent home with a commercial heart rate monitor. Participants will perform exercises at home on their free time 4-5 days per week. Participants will return to the clinic weekly to be re-examined by the study physician and obtain a new heart rate prescription for the first six weeks until clinical recovery or the intervention period ends (6-weeks).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40
* Received a concussion at work and are engaged with the workers compensation program
* Within 3 weeks of concussive injury

Exclusion Criteria:

* 3-point or less difference between current and pre-injury symptoms as measured by the Post-Concussion Symptom Inventory (PCSI)
* Moderate or severe TBI
* Injury involving loss of consciousness for >30 minutes or post-traumatic amnesia > 24 hours
* Pre-existing conditions or presence of polytrauma that prevent participation in active testing and/or rehabilitation
* History of more than 3 diagnosed concussions
* Active substance abuse/dependence
* Report of injury mechanism occurring due to physical assault
* Unwillingness to perform intervention
* Limited English proficiency.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Adherence to Target Heartrate Aerobic Exercise (THRAE) program as measured by counting the number and duration of exercise sessions completed. | Up to 6 weeks
  Adherence to Target Heartrate Aerobic Exercise (THRAE) program as measured by counting exercise sessions completed.

SECONDARY OUTCOMES:
Change in post-concussive symptom burden as measured by the Post-Concussion Symptom Scale | Baseline, week 1, week 2, week 3, week 4, week 5, week 6
  The Post-Concussion Symptom Scale (PCSS) is a validated 22-item self-report symptom questionnaire. Scores range from 0-132 with greater scores indicating increased symptom burden.
Change in Patient Health Questionnaire-9 (PHQ-9) | Baseline, up to week 6
  The Patient Health Questionnaire-9 (PHQ-9) is used for rating the severity of depression among participants. Scores range from 0-27. Higher scores indicate increased severity of depression.
Change in Generalized Anxiety Disorder-7 (GAD-7) | Baseline, up to week 6
  The Generalized Anxiety Disorder-7 (GAD-7) is used to measure the severity of anxiety among participants. Scores range from 0-21. Higher scores indicate increased severity of anxiety.
Primary Care Post Traumatic Stress Disorder (PTSD) Screen for DSM-5 (PC-PTSD-5) | Baseline
  The Primary Care Post Traumatic Stress Disorder (PTSD) Screen for DSM-5 (PC-PTSD-5) is used to measure probable PTSD among participants. Scores range from 0-5. Higher scores indicate increased probability of PTSD.
Change in Patient-Reported Outcomes Measurement Information System Global Health-10 (PROMIS-10) | Baseline, up to week 6
  The Patient-Reported Outcomes Measurement Information System Global Health-10 (PROMIS-10) is used to measure general healthcare-related quality of life, including global physical health and global mental health. Both global physical health and global mental health have raw scores ranging from 4-20. Higher scores reflect higher participant ratings for global physical and mental health. This measure will be used to assess change in global physical and mental health between the initial and final visits.
Work Climate Questionnaire - 6-Item Version | Baseline
  The Work Climate Questionnaire - 6-Item Version is used for assessing participants' perceptions regarding the degree of autonomy supportiveness of their work managers or employers. Scores range of 6-42. Higher scores indicate a greater degree of perceived autonomy supportiveness.
Change in Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS) | Baseline, up to week 6
  The Basic Psychological Needs Satisfaction and Frustration Scale (BPNSFS) is used to assess participant satisfaction or frustration with the psychological needs for autonomy, competence, and relatedness. The scale involves 6 subscales, including autonomy satisfaction, autonomy frustration, relatedness satisfaction, relatedness frustration, competence satisfaction, and competence frustration. Each subscale has scores ranging from 4-20. Higher scores indicate higher participant perceptions of the psychological need satisfaction or frustration reflected in the subscale. This measure will be used to assess change in psychological needs satisfaction and psychological needs frustration between the initial and final visits.
Time to return to work measured in days | Up to week 6
  Time to return to work as measured by difference between date of injury and date the participant is medically cleared to return to work

OTHER OUTCOMES:
Rate of adverse Events as assessed by questioning the participant | Up to week 6
  At each weekly follow-up meeting participants will be asked about any adverse events including injuries or other negative events.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob McPherson, Principal Investigator — SUNY Buffalo
Locations (1):
- UBMD Orthopaedics and Sports Medicine, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma B, Nowrouzi-Kia B, Mollayeva T, Kontos P, Grigorovich A, Liss G, Gibson B, Mantis S, Lewko J, Colantonio A. Work-related traumatic brain injury: A brief report on workers perspective on job and health and safety training, supervision, and injury preventability. Work. 2019;62(2):319-325. doi: 10.3233/WOR-192866. PMID 30829642
- [Background] Leddy JJ, Haider MN, Ellis MJ, Mannix R, Darling SR, Freitas MS, Suffoletto HN, Leiter J, Cordingley DM, Willer B. Early Subthreshold Aerobic Exercise for Sport-Related Concussion: A Randomized Clinical Trial. JAMA Pediatr. 2019 Apr 1;173(4):319-325. doi: 10.1001/jamapediatrics.2018.4397. PMID 30715132
- [Background] Leddy JJ, Master CL, Mannix R, Wiebe DJ, Grady MF, Meehan WP, Storey EP, Vernau BT, Brown NJ, Hunt D, Mohammed F, Mallon A, Rownd K, Arbogast KB, Cunningham A, Haider MN, Mayer AR, Willer BS. Early targeted heart rate aerobic exercise versus placebo stretching for sport-related concussion in adolescents: a randomised controlled trial. Lancet Child Adolesc Health. 2021 Nov;5(11):792-799. doi: 10.1016/S2352-4642(21)00267-4. Epub 2021 Oct 1. PMID 34600629
- [Background] de Koning ME, Scheenen ME, van der Horn HJ, Timmerman ME, Hageman G, Roks G, Spikman JM, van der Naalt J. Prediction of work resumption and sustainability up to 1 year after mild traumatic brain injury. Neurology. 2017 Oct 31;89(18):1908-1914. doi: 10.1212/WNL.0000000000004604. Epub 2017 Oct 6. PMID 28986414
- [Background] Kristman VL, Cote P, Van Eerd D, Vidmar M, Rezai M, Hogg-Johnson S, Wennberg RA, Cassidy JD. Prevalence of lost-time claims for mild traumatic brain injury in the working population: improving estimates using workers compensation databases. Brain Inj. 2008 Jan;22(1):51-9. doi: 10.1080/02699050701849991. PMID 18183509
- [Background] Smith CK, Wuellner S, Marcum J. Racial and ethnic disparities in workers' compensation claims rates. PLoS One. 2023 Jan 17;18(1):e0280307. doi: 10.1371/journal.pone.0280307. eCollection 2023. PMID 36649295
- [Derived] McPherson JI, Miecznikowski JC, Chizuk H, Sparks P, Leddy JJ, Haider MN, Stavisky CJ. Feasibility trial protocol assessing the use of aerobic exercise to promote recovery from work-related concussion. PLoS One. 2025 Jun 12;20(6):e0325701. doi: 10.1371/journal.pone.0325701. eCollection 2025. PMID 40504846

DOCUMENTS (1):
  • Informed Consent Form (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT06263179/ICF_000.pdf